CLINICAL TRIAL: NCT00326417
Title: Fludarabine-based Conditioning for Allogeneic Marrow Transplantation From HLA-compatible Unrelated Donors in Severe Aplastic Anemia (BMT CTN #0301)
Brief Title: Fludarabine-based Conditioning for Severe Aplastic Anemia (BMT CTN 0301)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN0301; U01HL069294 (NIH); 5U01HL069294-05 (NIH); 5U24CA076518 (NIH); NCT00335608 (obsolete NCT alias); NCT00474747 (obsolete NCT alias)
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Results first posted 2016-10-04 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Anemia, Aplastic
Keywords: Severe Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cyclophosphamide 150mg (Experimental): Fludarabine plus 150 mg/kg Cyclophosphamide (total dose)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide 150mg
- Cyclophosphamide 100mg (Experimental): Fludarabine plus 100 mg/kg Cyclophosphamide (total dose)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide 100mg
- Cyclophosphamide 50mg (Experimental): Fludarabine plus 50 mg/kg Cyclophosphamide (total dose)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide 50mg
- Fludarabine (Experimental): Fludarabine only (no Cyclophosphamide administered)
  Interventions: Drug: Fludarabine

INTERVENTIONS:
Drug: Fludarabine — Doses of 30 mg/m^2 IV will be given for no less than 30 minutes daily for 4 days (Days -5 to -2)
  Other Names: Fludara
Drug: Cyclophosphamide 150mg — A total dose of 150 mg/kg will be given as 50 mg/kg per day for 3 days (Days -4, -3, -2)
  Other Names: Cytoxan®
  Arms: Cyclophosphamide 150mg
Drug: Cyclophosphamide 100mg — A total dose of 100 mg/kg will be given as 50 mg/kg per day for 2 days (Days -3, -2)
  Other Names: Cytoxan®
  Arms: Cyclophosphamide 100mg
Drug: Cyclophosphamide 50mg — A total dose of 50 mg/kg will be given once at 50 mg/kg per day on Day -2
  Other Names: Cytoxan®
  Arms: Cyclophosphamide 50mg

SUMMARY:
The purpose of the current study is to continue to optimize conditioning regimens in high-risk patients with severe aplastic anemia transplanted with marrow from HLA-compatible unrelated donors. Specifically, the study will determine whether the addition of fludarabine to the conditioning regimen previously described by Deeg et al. will permit a reduction in the CY dose, to a point where sustained hematopoietic engraftment and survival are maintained (or improved), while the frequency of major regimen-related toxicity (RRT) and early deaths is reduced.

DETAILED DESCRIPTION:
BACKGROUND:

Aplastic anemia (AA) remains a life-threatening illness. Treatment options include supportive care (transfusions, growth factors, etc.), immunosuppression therapy and stem cell transplantation. Only the latter two have favorably impacted the natural history of the disease. The prognosis of AA patients, particularly severe aplastic anemia (SAA), as defined by Camitta et al., who fail to respond to immunosuppressive therapy (IS) or who relapse after an initial response to IS is poor. Although many of these patients can be supported in the short term with growth factors, transfusions and possibly rechallenged successfully with IS, the cumulative morbidity and mortality from infection, hemorrhage or transfusion-related complications is substantial.

While allogeneic bone marrow transplantation is potentially curative in AA, no more than 25% of patients have a human leukocyte antigen (HLA)-identical sibling donor. Cyclophosphamide (CY)-antithymocyte globulin (ATG) has been recommended as the preparative regimen of choice in sibling donor transplants. Results of bone marrow transplantation from alternative donors, such as matched unrelated donors and mismatched related donors in AA patients who have failed IS, have largely been unsatisfactory. The cyclophosphamide-ATG conditioning regimen has proved inadequate in ensuring engraftment in allogeneic transplants from matched, unrelated donors for AA. This was the major reason why total body radiation (TBI) has been added to the conditioning regimen.

Graft failure is a very serious and frequently life-threatening or fatal event following matched unrelated donor (MUD) allografts in aplastic anemia. It is an immunologically mediated event. Risk factors for graft failure include the use of HLA nonidentical or unrelated donors, a poor marrow nucleated cell dose as well as prolonged transfusional support prior to BMT (which increases the probability of patient sensitization to multiple antigens). While some patients may achieve autologous hematopoietic recovery, prolonged pancytopenia is common and infection-related morbidity and mortality are very substantial. Reconditioning for a second allograft from the same or a different donor is frequently not successful. While the addition of TBI and intensive pre-transplant conditioning has led to a sizable improvement in engraftment rates, this has come with a price, particularly in adult patients. Transplant-related toxicity has been a major and frequent problem. Radiation-induced pulmonary toxicity in particular has been common, usually in the form of diffuse alveolar damage or diffuse interstitial pneumonitis. In addition, Graft Versus Host Disease (GVHD)-related morbidity and mortality in these patients have also been substantial.

DESIGN NARRATIVE:

The study is a prospective Phase I/II dose optimization study. All patients are given a fixed dose of ATG (either thymoglobulin: 3 mg/kg IV daily x 3 or ATGAM 30 mg/kg IV daily x 3, on Days -4 to -2), Fludarabine (30 mg/m^2 IV daily x 4, on Days - 5 to -2), and TBI (200 cGy (centigray) from a linear accelerator at less than 20 cGy/min on Day -1). The starting CY dose will be 150 mg/kg (50 mg/kg intravenously daily, Days -4 to -2), and will be de-escalated depending on engraftment and toxicity. The Phase I portion of the trial (maximum of 24-27 patients) tests each of four dose levels of CY for adequate safety and graft retention. The Phase II portion of the trial refines the dose selection and allocates an additional 70 patients to the optimal dose, at which two-year post-transplant survival will be assessed. The combined enrollment in Phase I and II will total 94 patients.

The study is a prospective single-arm Phase I/II dose-selection and evaluation study. The study will seek the optimal dose level of CY based on assessments of graft failure, toxicity and early death during 100 days of follow-up post-transplant. A brief synopsis is given below.

Phase I - Test Each Dose for Adequate Safety and Graft Retention

1. Proceed from the highest dose (150 mg/kg CY) to the lowest dose (0 mg/kg CY), treating a minimum of six patients at each dose.
2. Evaluate the 100-Day outcomes for toxicity, death and graft failure on each patient enrolled at the current dose, or until stopping criteria are met.
3. If there are three or more graft failures at the current dose, the current dose and all lower doses are closed to further enrollment.
4. If there are five or more severe regimen-related toxicities and/or early deaths at the current dose, the current dose is closed to further enrollment, and the next lower dose is tested.
5. Dose de-escalation ceases once all four doses are tested or closed to further enrollment.

Phase II - Refine Dose Selection and Allocate Patients to the Optimal Dose

1. Treat each newly enrolled patient at the most desirable of the dose levels remaining open to enrollment. This can involve de-escalation, escalation, or no change in dose.
2. As each patient completes the observation period, evaluate the 100-Day outcomes for graft failure, toxicity and/or early death for this patient, or until stopping criteria are met.
3. If there are excess (according to the criteria in Table 5.8) graft failures, that patient's dose and all lower doses are closed to further enrollment.
4. If there are excess (according to the criteria in Table 5.8) toxicities and/or early deaths, that patient's dose is closed to further enrollment.
5. Re-evaluate the desirability of the current dose level based on the 100-Day outcomes for toxicity and/or early death and graft failure.
6. Repeat steps 1-5 until 54 patients are enrolled in Phase II, or all dose levels are closed to further enrollment.

Dosage Levels for CY:

3 Days (Day -4, -3, -2): Dose of 50 mg/kg/day; total dose of 150 mg/kg; dose level 3

2 Days (Day -3, -2): Dose of 50 mg/kg/day; total dose of 100 mg/kg; dose level 2

1 Day (Day -2): Dose of 50 mg/kg/day; total dose of 50 mg/kg; dose level 1

0 Days (None): No dose; no total dose; dose level 0

There may be wait periods between enrollment of successive patients and/or cohorts for endpoint assessment. Under these circumstances, the final decision about waiting versus treating the patient off study will be made at the local transplant center.

ELIGIBILITY:
Inclusion Criteria:

* Patients up to 65 years of age at time of registration with a diagnosis of SAA; SAA is defined as follows:

  1. Bone marrow cellularity less than 25% or marrow cellularity less than 50% but with less than 30% residual hematopoietic cells
  2. Two out of three of the following (in peripheral blood): neutrophils less than 0.5 x 10^9/L; platelets less than 20 x 10^9/L; reticulocytes less than 20 x 10^9/L
* Patient must have an available unrelated donor with a 7/8 or 8/8 match for HLA-A, B, C, and DRB1 antigen; typing is by DNA techniques: intermediate resolution for A, B, and C, and high resolution for DRB1; HLA-DQ typing is recommended but will not count in the match
* Patient and/or legal guardian able to provide signed informed consent
* Matched unrelated donor must consent to provide a marrow allograft
* Patients with adequate organ function as measured by:

  1. Cardiac: left ventricular ejection fraction at rest must be greater than 40% or shortening fraction greater than 20%
  2. Hepatic: serum bilirubin less than 2x upper limit of normal for age as per local laboratory) (with the exception of isolated hyperbilirubinemia due to Gilbert's syndrome), alanine transaminase (ALT) and aspartate transaminase (AST) less than 4x upper limit of normal for age (as per local laboratory)
  3. Renal: serum creatinine less than 2x upper limit of normal for age (as per local laboratory)
  4. Pulmonary: Forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), and carbon monoxide diffusing capacity (DLCO) (corrected for Hb) greater than 50% predicted; for patients in which pulse oxymetry is performed, O2 saturation greater than 92%
* Diagnosis of Fanconi anemia must be excluded in patients younger than 18 years of age by diepoxybutane testing on peripheral blood or comparable testing on marrow.

Exclusion Criteria:

* Clonal cytogenetic abnormalities associated with myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) on marrow examination
* Diagnosis of other "congenital" aplastic anemias such as: Diamond-Blackfan; Shwachman-Diamond; congenital amegakaryocytosis
* Symptomatic or uncontrolled cardiac failure or coronary artery disease
* Karnofsky performance status less than 60% or Lansky less than 40% for patients younger than 16 years old
* Uncontrolled bacterial, viral or fungal infections (currently taking medication and progression of clinical symptoms)
* Seropositive for the human immunodeficiency virus (HIV)
* Pregnant (positive total HCG) or breastfeeding
* Presence of large accumulation of ascites or pleural effusions, which would be a contraindication to the administration of methotrexate for GVHD prophylaxis
* Known severe or life-threatening allergy or intolerance to ATG or cyclosporine/ tacrolimus
* Planned administration of alemtuzumab (Campath-1H) or other investigational agents as alternative agent for GVHD prophylaxis
* Concomitant enrollment in a Phase I study
* Positive patient anti-donor lymphocyte crossmatch in HLA-A or B mismatched transplants; the definition of match is in Section 2.2.1; the crossmatch would only apply to mismatches at HLA-A or B, not DRB1 or HLA-C
* Prior allogeneic marrow or stem cell transplantation
* Patients with prior malignancies except resected basal cell carcinoma or treated carcinoma in-situ; cancer treated with curative intent less than 5 years previously will not be allowed unless approved by the Medical Monitor or Protocol Chair; cancer treated with curative intent more than 5 years previously will be allowed

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2006-01; Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (22):
- United States (22):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital at UCLA, Los Angeles, California
  - Stanford Hospital and Clinics, Stanford, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - BMT Program at Northside Hospital, Atlanta, Georgia
  - DFCI/Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Texas, MD Anderson CRC, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Virginia Commonwealth University, MCV Hospital, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Findings will be published in a manuscript.
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public.
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Background] Pulsipher MA, Young NS, Tolar J, Risitano AM, Deeg HJ, Anderlini P, Calado R, Kojima S, Eapen M, Harris R, Scheinberg P, Savage S, Maciejewski JP, Tiu RV, DiFronzo N, Horowitz MM, Antin JH. Optimization of therapy for severe aplastic anemia based on clinical, biologic, and treatment response parameters: conclusions of an international working group on severe aplastic anemia convened by the Blood and Marrow Transplant Clinical Trials Network, March 2010. Biol Blood Marrow Transplant. 2011 Mar;17(3):291-9. doi: 10.1016/j.bbmt.2010.10.028. Epub 2010 Oct 27. PMID 21034841
- [Result] Anderlini P, Wu J, Gersten I, Ewell M, Tolar J, Antin JH, Adams R, Arai S, Eames G, Horwitz ME, McCarty J, Nakamura R, Pulsipher MA, Rowley S, Leifer E, Carter SL, DiFronzo NL, Horowitz MM, Confer D, Deeg HJ, Eapen M. Cyclophosphamide conditioning in patients with severe aplastic anaemia given unrelated marrow transplantation: a phase 1-2 dose de-escalation study. Lancet Haematol. 2015 Sep;2(9):e367-75. doi: 10.1016/S2352-3026(15)00147-7. Epub 2015 Sep 2. PMID 26685770
- [Result] Tolar J, Deeg HJ, Arai S, Horwitz M, Antin JH, McCarty JM, Adams RH, Ewell M, Leifer ES, Gersten ID, Carter SL, Horowitz MM, Nakamura R, Pulsipher MA, Difronzo NL, Confer DL, Eapen M, Anderlini P. Fludarabine-based conditioning for marrow transplantation from unrelated donors in severe aplastic anemia: early results of a cyclophosphamide dose deescalation study show life-threatening adverse events at predefined cyclophosphamide dose levels. Biol Blood Marrow Transplant. 2012 Jul;18(7):1007-11. doi: 10.1016/j.bbmt.2012.04.014. Epub 2012 Apr 27. PMID 22546497

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from February 2006 to August 2007 for Phase I of the trial. Phase II opened in November 2007 and closed to accrual on December 2, 2013.
Period: Overall Study
Arm/Group | Cyclophosphamide 150mg | Cyclophosphamide 100mg | Cyclophosphamide 50mg | Fludarabine
Started | 14 | 41 | 39 | 3
Phase I | 6 | 6 | 6 | 3
Phase II | 8 | 35 | 33 | 0
Completed | 0 (Dose level was closed for excessive toxicity after 8 patients in Phase II accrued.) | 41 | 38 | 0 (Arm was closed to accrual after 3 patients experienced graft failure.)
Not Completed | 14 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Arm Closed | 7 | 0 | 0 | 3
Not completed — Death | 7 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclophosphamide 100mg | Cyclophosphamide 50mg | Total
Number analyzed (Participants) | 41 | 38 | 79
Age, Continuous [Median (Full Range); unit: years] | 17.6 [1.9 to 63.3] | 24.5 [0.5 to 65.9] | 20.6 [0.5 to 65.9]
Age, Customized [Number; unit: participants]
  < 18 | 21 | 11 | 32
  18 - 40 | 14 | 18 | 32
  > 40 | 6 | 9 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 21 | 19 | 40
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 34 | 30 | 64
  Hispanic or Latino | 6 | 8 | 14
  Unknown | 1 | 0 | 1
Recipient Cytomegalovirus Status [Number; unit: participants]
  Positive | 26 | 17 | 43
  Negative | 15 | 21 | 36
Karnofsky Score [Number; unit: participants] — Assesses patient self-perceived global quality of life and functioning (excellent, very good, good, fair, poor), where 100 equals perfect quality of life.
  participants
    100 | 18 | 12 | 30
    90 | 15 | 17 | 32
    80 | 3 | 7 | 10
    70 | 4 | 2 | 6
    60 | 1 | 0 | 1
Immunosuppressive therapy prior to transplant [Number; unit: participants]
  Yes | 41 | 35 | 76
  No | 0 | 3 | 3
Donor-recipient HLA match [Number; unit: participants]
  HLA-A, -B, -C,-DRB1 matched | 27 | 31 | 58
  Single HLA-locus mismatch | 14 | 7 | 21
Type of anti-thymocyte globulin administered [Number; unit: participants]
  Rabbit-derived | 33 | 29 | 62
  Horse-derived | 7 | 9 | 16
  None | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)
Description: DFS includes graft failure, regimen-related toxicity (RRT), and early death. Graft Failure is defined by lack of neutrophil engraftment (ANC less than 0.5 x 10^9/L for 3 consecutive days on different days). Major RRT is defined as severity of grade 4 in any organ system or grade 3 for pulmonary, cardiac, renal, oral mucosal or hepatic. Early death is defined as death prior to Day 100 post-transplant.
Time Frame: Day 100
Measure: Number; unit: participants
Arm/Group | Cyclophosphamide 100mg | Cyclophosphamide 50mg
Number analyzed (Participants) | 41 | 38
participants
  Graft Failure | 6 | 3
  Major RRT | 9 | 4
  Survival | 39 | 37
  Alive and engrafted | 35 | 35

2. Secondary Outcome: Cumulative Incidence of Graft Failure
Description: Primary and secondary graft failure are included, secondary graft failure is defined by initial neutrophil engraftment followed by subsequent decline in the ANC to less than 0.5 x 10^9/L for three consecutive measurements on different days, unresponsive to growth factor.
Time Frame: Day 365
Measure: Number; unit: percentage of participants
Arm/Group | Cyclophosphamide 100mg | Cyclophosphamide 50mg
Number analyzed (Participants) | 41 | 38
percentage of participants | 14.6 | 11.7

3. Secondary Outcome: Acute Graft vs Host Disease (GVHD)
Description: All GVHD grades 2-4 will be graded according to the BMT CTN Manual of Procedures (MOP)
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclophosphamide 100mg | Cyclophosphamide 50mg
Number analyzed (Participants) | 41 | 38
percentage of participants | 26.8 [13 to 40.6] | 23.7 [10 to 37.4]

4. Secondary Outcome: Chronic GVHD
Description: Chronic GVHD is scored according to the BMT CTN MOP. The first day of chronic GVHD onset will be used to calculate cumulative incidence curves.
Time Frame: Day 365
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclophosphamide 100mg | Cyclophosphamide 50mg
Number analyzed (Participants) | 41 | 38
percentage of participants | 31.7 [18.1 to 46.2] | 22.5 [10.3 to 37.5]

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as alive at 1 year, the event is death from any cause. Patients alive at the time of last observation, for statistical purposes, will have a survival time which is censored.
Time Frame: Day 365
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclophosphamide 100mg | Cyclophosphamide 50mg
Number analyzed (Participants) | 41 | 38
percentage of participants | 80.5 [64.8 to 89.7] | 97.4 [82.8 to 99.6]

ADVERSE EVENTS:
Time Frame: 1 year post-transplant
Description: Serious Adverse Events (AE) are defined as events associated with death, life-threatening event, disability, congenital anomaly, required intervention to prevent permanent impairment or damage, hospitalization or other serious adverse event. Only unexpected grades 3-5 adverse events were required to be reported through the AE system per protocol.
Arm/Group | Cyclophosphamide 150mg | Cyclophosphamide 100mg | Cyclophosphamide 50mg | Fludarabine
Serious Adverse Events (participants affected / at risk) | 8/14 | 4/41 | 4/38 | 1/3
Other Adverse Events (participants affected / at risk) | 0/14 | 1/41 | 0/38 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide 150mg (N=14) | Cyclophosphamide 100mg (N=41) | Cyclophosphamide 50mg (N=38) | Fludarabine (N=3)
Papilloedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 7 (7) | 2 (2) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide 150mg (N=14) | Cyclophosphamide 100mg (N=41) | Cyclophosphamide 50mg (N=38) | Fludarabine (N=3)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-06-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT00326417/Prot_SAP_ICF_000.pdf